CLINICAL TRIAL: NCT02467452
Title: A Multinational, Multicentre, Randomised, Open-Label, Active-Controlled, 26-Week, 2-Arm, Parallel Group Study to Evaluate the Non-Inferiority of Fixed Combination of Beclomethasone Dipropionate Plus Formoterol Fumarate Plus Glycopyrronium Bromide (CHF 5993) Administered Via Pressurized Metered-dose Inhaler (pMDI) Versus Fixed Combination Of Fluticasone Furoate Plus Vilanterol Administered Via Dry Powder Inhaler (DPI) (Relvar®) Plus Tiotropium Bromide (Spiriva®) for the Treatment of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Non Inferiority of Fixed Combination of Beclomethasone Dipropionate (BDP) + Formoterol Fumarate (FF) + Glycopyrronium Bromide (GB) Versus Combination of Fluticasone Furoate (FlF)/Vilanterol (VI) + Tiotropium Bromide in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCD-05993AA1-07; 2014-001487-35 (EudraCT Number)
Record Dates: First submitted 2015-05-20; First posted 2015-06-10 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BDP/FF/GB (Experimental): Drug: BDP/FF/GB Other name: CHF 5993 pMDI 100/6/12 mcg
  Interventions: Drug: BDP/FF/GB
- FlF/VI + Tiotropium (Active Comparator): FlF/VI + Tiotropium Other name: Relvar DPI 100/25 mcg + Spiriva 18 mcg capsule
  Interventions: Drug: FlF/VI + Tiotropium

INTERVENTIONS:
Drug: BDP/FF/GB
  Arms: BDP/FF/GB
Drug: FlF/VI + Tiotropium
  Arms: FlF/VI + Tiotropium

SUMMARY:
The purpose of the study is to demonstrate the triple combination of beclometasone dipropionate + formoterol fumarate + glycopyrronium bromide is effective in term of quality of life in COPD patients (Chronic Obstructive Pulmonary Disease).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged ≥ 40 years with written informed consent obtained prior to any study-related procedure.
2. Patients with a diagnosis of COPD at least 12 months before the screening visit (according to GOLD document updated 2014).
3. Current smokers or ex-smokers who quit smoking at least 6 months prior to screening visit, with a smoking history of at least 10 pack years [pack-years = (number of cigarettes per day x number of years)/20].
4. A post-bronchodilator FEV1 < 50% of the predicted normal value and a post-bronchodilator forced expiratory volume at one second (FEV1)/forced vital capacity (FVC) < 0.7 at least 10-15 min after 4 puffs (4 x 100 μg) of salbutamol pMDI. If this criterion is not met at screening, the test can be repeated once before randomisation.
5. A documented history of at least one exacerbation in the 12 months preceding the screening visit.

   COPD exacerbation will be defined according to the following:

   "A sustained worsening of the patient's condition (dyspnoea, cough and/or sputum production/purulence), from the stable state and beyond normal day-to-day variations, that is acute in onset and necessitates a change in regular medication in a patient with underlying COPD that includes prescriptions of systemic corticosteroids and/or antibiotics or need for hospitalization". Also documented visits to an emergency department due to COPD exacerbation are considered acceptable to fulfil this criterion.
6. Patients under double therapy for at least 2 months prior to screening visit with either:

   1. inhaled corticosteroids/long-acting β2-agonist combination (fixed or free), without regular use of short-acting muscarinic antagonist (regular use means 2 puffs 4 times per day at least) or
   2. inhaled corticosteroids/long-acting muscarinic antagonist free combination, without regular use of short-acting β2-agonist (regular use means 2 puffs 4 times per day at least) or
   3. Inhaled long-acting β2-agonist and inhaled long-acting muscarinic antagonist or
   4. Patients under monotherapy with long-acting muscarinic antagonist for at least 2 months prior to screening.
7. Symptomatic patients at screening with a CAT score ≥10.
8. A cooperative attitude and ability to use correctly the inhalers.
9. A cooperative attitude and ability to use correctly the daily electronic Diary (eDiary).

Exclusion Criteria:

1. Pregnant or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential) UNLESS are willing to use one or more methods of contraception as defined in the protocol
2. Patients with a current clinical diagnosis of asthma with a physician-judged need for inhaled or oral corticosteroid therapy
3. Patients requiring use of the following medications:

   1. A course of systemic steroids longer than 3 days for COPD exacerbation in the 4 weeks prior to screening
   2. A course of antibiotics for COPD exacerbation longer than 7 days in the 4 weeks prior to screening
   3. phosphodiesterase-4 (PDE4) inhibitors in the 4 weeks prior to screening
   4. Use of antibiotics for a lower respiratory tract infection (e.g pneumonia) in the 4 weeks prior to screening
4. COPD exacerbation requiring prescriptions of systemic corticosteroids and/or antibiotics or hospitalization during the run-in period
5. Patients treated with non-cardio selective β-blockers in the month preceding the screening visit or during the run-in period. Those patients may enter the study after non-selective β-blockers withdrawal and/or cardio selective β-blockers intake for at least 10 days before randomization
6. Patients treated with long-acting antihistamines unless taken at stable regimen at least 2 months prior to screening and to be maintained constant during the study, or if taken as o re nata (PRN).
7. Patients requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia.
8. Known respiratory disorders other than COPD which may impact the efficacy of the study drug according the investigator's judgment
9. Patients who have clinically significant cardiovascular condition
10. Patients with atrial fibrillation (AF):

    1. Paroxysmal Atrial Fibrillation
    2. Persistent: AF episode either lasts longer than 7 days or requires termination by cardioversion, either with drugs or by direct current cardioversion (DCC) within 6 months from screening
    3. Long standing Persistent as defined by continuous atrial fibrillation diagnosed for less than 6 months with or without a rhythm control strategy
    4. Permanent: for at least 6 months with a resting ventricular rate ≥ 100/min controlled with a rate control strategy (i.e., selective β-blocker, calcium channel blocker, pacemaker placement, digoxin or ablation therapy)
11. An abnormal and clinically significant 12-lead ECG which may impact the safety of the patient according to investigator's judgement Patients whose electrocardiogram (ECG12 lead) shows QT Interval Corrected by the Fridericia Correction Formula (QTcF) >450 ms for males or QTcF >470 ms for females at screening visit are not eligible (not applicable for patient with pacemaker)
12. Medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the investigator would prevent use of anticholinergic agents
13. History of hypersensitivity to anticholinergics, β2-agonist, corticosteroids or any of the excipients contained in any of the formulations used in the trial which may raise contra-indications or impact the efficacy of the study drug according to the investigator's judgement
14. Clinically significant laboratory abnormalities indicating a significant or unstable concomitant disease which may impact the efficacy or the safety of the study drug according to investigator's judgement
15. Patients with hypokalaemia (serum potassium levels <3.5 milliequivalent per liter (mEq/L) (or 3.5 mmol/L)) or uncontrolled hyperkalaemia according to investigator's judgment
16. Unstable concurrent disease: e.g. uncontrolled hyperthyroidism, uncontrolled diabetes mellitus or other endocrine disease; significant hepatic impairment; significant renal impairment; uncontrolled gastrointestinal disease (e.g. active peptic ulcer); uncontrolled neurological disease; uncontrolled haematological disease; uncontrolled autoimmune disorders, or other which may impact the efficacy or the safety of the study drug according to investigator's judgment.
17. Patients with any history of malignancy likely to result in significant disability or likely to require significant medical or surgical intervention within the next six months (after V1) or with malignancy for which they are currently undergoing radiation therapy or chemotherapy
18. History of alcohol abuse and/or substance/drug abuse within 12 months prior to screening visit
19. Participation in another clinical trial where investigation drug was received less than 8 weeks prior to screening visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1479 (Actual)
Dates: Start 2015-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Saint George's Respiratory Questionnaire (SGRQ) total score at Week 26. | 26 weeks
  the primary efficacy variable is the numeric value of the change

SECONDARY OUTCOMES:
SGRQ response (change from baseline in total score ≤ -4) at Week 26. | 26 weeks
  the secondary efficacy variable is derived as a categorisation of this value
rced expiratory volume at one second (FEV1) response (change from baseline in pre-dose morning FEV1 ≥ 100 ml) at Week 26. | 26 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Erzsebet Gondozohaz, Gödöllő, Hungary

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2014-001487-35/results
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/15_CSR_Synopsis_CCD-05993AA1-07.pdf